CLINICAL TRIAL: NCT01901094
Title: A Randomized Phase III Trial Comparing Axillary Lymph Node Dissection to Axillary Radiation in Breast Cancer Patients (cT1-3 N1) Who Have Positive Sentinel Lymph Node Disease After Neoadjuvant Chemotherapy
Brief Title: Comparison of Axillary Lymph Node Dissection with Axillary Radiation for Patients with Node-Positive Breast Cancer Treated with Chemotherapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A011202; U10CA031946 (NIH); NCI-2013-00875 (Registry Identifier: Clinical Trial Reporting Program)
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Stage II Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: ALND + nodal radiation therapy (Other): Surgery: For patients randomized to axillary lymph node dissection (ALND), it is recommended that a complete level I and II dissection with resection of minimum of a total of 8 lymph nodes (SLN and ALND together) be done. Level III dissection is not required, but may be performed at the discretion of the surgeon. If fewer than 8 lymph nodes (SLN and ALND together) are resected, then the patient will discontinue protocol treatment.
  Radiation Therapy: Radiation is delivered to the breast/chest wall, undissected axilla, supraclavicular nodes and internal mammary nodes in the first 3 intercostal spaces. Treatment will be given 5 days a week over 5-6 weeks.
  Interventions: Procedure: Axillary Lymph Node Dissection (ALND); Radiation: Nodal Radiation Therapy
- Arm 2: Axillary radiation and nodal radiation therapy (Other): Radiation Therapy: Radiation is delivered to the breast/chest wall, full axilla including Levels I, II, III, supraclavicular nodes and internal mammary nodes in the first 3 intercostal spaces. Treatment will be given 5 days a week over 5-6 weeks.
  Interventions: Radiation: Nodal Radiation Therapy; Radiation: Axillary Radiation Therapy

INTERVENTIONS:
Procedure: Axillary Lymph Node Dissection (ALND)
  Arms: Arm 1: ALND + nodal radiation therapy
Radiation: Nodal Radiation Therapy
Radiation: Axillary Radiation Therapy
  Arms: Arm 2: Axillary radiation and nodal radiation therapy

SUMMARY:
This randomized phase III trial studies lymph node dissection and radiation therapy to see how well it works compared to radiation therapy alone in treating patients with breast cancer previously treated with chemotherapy and surgery. Lymph node dissection may remove cancer cells that have spread to nearby lymph nodes in patients with breast cancer. Radiation therapy uses high-energy x rays or protons to kill tumor cells. It is not yet known if radiation therapy works better alone or with lymph node dissection in treating patients with breast cancer previously treated with chemotherapy and surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether radiation to the undissected axilla and regional lymph nodes is not inferior to axillary lymph node dissection with radiation to the regional lymph nodes but not to the dissected axilla in terms of invasive breast cancer recurrence-free interval in patients with positive sentinel lymph node(s) (SLN[s]) after completion of neoadjuvant chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate whether radiation to the undissected axilla and regional lymph nodes is not inferior to axillary lymph node dissection with radiation to the regional lymph nodes but not to the dissected axilla in terms of the incidence of invasive loco-regional recurrences in patients with a positive SLN(s) after completion of neoadjuvant chemotherapy.

II. To obtain an estimate of the distribution of residual disease burden scores.

III. To estimate the distribution of overall survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo axillary lymph node dissection. Beginning 3-12 weeks following surgery, patients undergo nodal radiation therapy comprising 3-dimensional (3D) conformal radiation therapy (3D-CRT), intensity-modulated radiation therapy (IMRT), or proton radiation therapy (PRT) 5 days a week for 5-6 weeks.

ARM II: Patients undergo axillary and nodal radiation therapy comprising 3D-CRT, IMRT, or PRT 5 days a week for 5-6 weeks.

After completion of study treatment, patients are followed up at least every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Pre-Registration Eligibility Criteria:

* Clinical stage T1-3 N1 M0 breast cancer at diagnosis (prior to the start of neoadjuvant chemotherapy) by American Joint Committee on Cancer (AJCC) staging 7th edition
* No inflammatory breast cancer
* No other malignancy within 5 years of registration with the exception of basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the cervix
* All patients must have had an axillary ultrasound with fine needle aspiration (FNA) or core needle biopsy of axillary lymph nodes documenting axillary metastasis at the time of diagnosis, prior to or at most 14 days after starting neoadjuvant chemotherapy

  * Note: Biopsy of intramammary nodes does not fulfill eligibility criteria
* Patients must have had estrogen receptor, progesterone receptor and HER2 status (by immunohistochemistry [IHC] and/or in situ hybridization [ISH]) evaluated on diagnostic core biopsy prior to start of neoadjuvant chemotherapy

  * Note: If HER2 status has not been clearly determined (i.e. equivocal/indeterminate), then patients should not be enrolled
* Patients must have completed all planned neoadjuvant chemotherapy prior to surgery; sandwich chemotherapy is not allowed (i.e. anthracycline/cytoxan or taxane chemotherapy planned to be given after surgery); patients must have completed at least 4 cycles of neoadjuvant chemotherapy consisting of an anthracycline and/or taxane-based regimen without evidence of disease progression in the breast or the lymph nodes

  * Note: Delays/dose modifications due to toxicities/adverse events are allowed as long as a minimum of 4 cycles of neoadjuvant chemotherapy is administered; more than 4 cycles of neoadjuvant chemotherapy (NAC) may be administered at the discretion of the treating medical oncologist
* Patients with HER-2 positive tumors must have received neoadjuvant trastuzumab, or trastuzumab + pertuzumab, or other approved anti-HER-2 therapy (either with all or with a portion of the neoadjuvant chemotherapy regimen); therapy must be Food and Drug Administration (FDA)-approved targeted anti-HER2 therapy, but additional therapies are allowed as are non-trastuzumab regimens if administered in the context of an Institutional Review Board (IRB)-approved clinical trial
* All patients must have a clinically negative axilla (no bulky adenopathy) on physical examination documented at the completion of neoadjuvant chemotherapy

  * Note: an ultrasound of the axilla is not required at completion of neoadjuvant chemotherapy; if performed, its findings do NOT impact eligibility
* No more than 8 weeks of neoadjuvant endocrine therapy prior to the start of neoadjuvant chemotherapy
* No neoadjuvant radiation therapy
* No SLN surgery/excisional biopsy for pathological confirmation of axillary status prior to or during neoadjuvant chemotherapy
* No prior history of ipsilateral breast cancer (invasive disease or ductal carcinoma in situ [DCIS]); lobular carcinoma in situ (LCIS) and benign breast disease is allowed
* No prior ipsilateral axillary surgery, such as excisional biopsy of lymph node(s) or treatment of hidradenitis
* No history of prior or concurrent contralateral invasive breast cancer; benign breast disease; LCIS or DCIS of contralateral breast is allowed
* Patients must not be pregnant or nursing

  * Note: Peri-menopausal women must be amenorrheic for > 12 months to be considered not of childbearing potential
* Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status 0-1

Intra-Operative Registration/Randomization Criteria:

* Breast surgery (lumpectomy or mastectomy) and sentinel lymph node surgery must be completed within 56 days of the completion of the last dose of neoadjuvant chemotherapy
* A minimum of 1 sentinel node and a maximum of 8 total nodes (sentinel + non-sentinel) are identified and excised; more than 8 nodes identified by either surgeon or pathologist is NOT allowed Note: Patients who do not have an identifiable sentinel lymph node will not proceed to registration/randomization
* At least one lymph node (sentinel or non-sentinel) excised during sentinel lymph node surgery with a metastasis greater than 0.2 mm in greatest dimension identified on intra-operative pathologic assessment

  * Note: Isolated tumor cells (metastases less than or equal to 0.2 mm) will be treated as node negative disease (N0i+)
  * Note: If on final pathology, more than 8 lymph nodes are seen pathologically, then the patient should discontinue study
  * Axillary lymph node dissection (ALND) is not to be performed prior to registration/randomization
  * Note: Patients for whom no positive lymph nodes (sentinel or non-sentinel) are found during sentinel lymph node surgery will not proceed to registration/randomization and can be considered for discussion of the NRG NSABP B-51/RTOG 1304 study "A Randomized Phase III Clinical Trial Evaluating the Role of Post-mastectomy Chest Wall and Regional Nodal XRT and Post-lumpectomy Regional Nodal XRT in Patients with Documented Positive Axillary Nodes Before Neoadjuvant Chemotherapy Who Convert to Pathologically Negative Axillary Nodes After Neoadjuvant Chemotherapy"

Post-Operative Registration/Randomization Criteria:

* For cases where ALND has not been performed and one of the following is true: 1) intra-operative evaluation of sentinel lymph node could not be/was not performed and final pathology identified a positive lymph node (sentinel or non-sentinel) with metastasis greater than 0.2 mm OR 2) lymph node (sentinel or non-sentinel) considered negative on intra-operative evaluation was found to be positive on final pathology (with metastasis greater than 0.2 mm)
* Breast surgery (lumpectomy or mastectomy) and sentinel lymph node surgery must be completed within 56 days of the completion of the last dose of neoadjuvant chemotherapy; negative margin (by either breast conservation or mastectomy) on final pathology where negative margin is defined as no tumor on ink
* At least one lymph node (sentinel or non-sentinel) with a metastasis greater than 0.2 mm in greatest dimension identified on final pathology (for cases where intra-operative evaluation was not performed, or was negative and completion dissection was not performed)
* At least one and no more than 8 lymph nodes (sentinel and non-sentinel) were found by the pathologists to have been actually excised during sentinel lymph node procedure Note: Isolated tumor cells (metastases less than or equal to 0.2 mm) will be treated as node negative disease (N0i+)
* For those patients who also undergo contralateral breast surgery, if invasive disease is found in the contralateral breast, the patient is not eligible for registration /randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2012 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Invasive breast cancer recurrence-free interval (IBC-RFI) | Up to 8 years after completion of radiation therapy

SECONDARY OUTCOMES:
Overall survival | Up to 8 years after completion of radiation therapy
Ipsilateral/local/regional invasive breast cancer recurrence (ILR-REC) | Up to 8 years after completion of radiation therapy

OTHER OUTCOMES:
Development of arm lymphedema if there is a 10% increase in the volume of the ipsilateral arm from its pre-surgery volume | Up to 5 years after completion of radiation therapy
Breast lymphedema (in BCT patients) | Up to 5 years after completion of radiation therapy
Adequacy of radiation fields, dose delivered to supraclavicular and axillary nodes | Up to 8 years after completion of radiation therapy
Residual cancer burden (RCB) | Up to 8 years after completion of radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Judy Boughey, MD, Study Chair — Mayo Clinic
Locations (1246):
- United States (1228):
  - Southern Cancer Center PC-Daphne, Daphne, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Southern Cancer Center PC-Mobile, Mobile, Alabama
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Southern Cancer Center PC-Springhill, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arizona Breast Cancer Specialists-Gilbert, Gilbert, Arizona
  - Virginia G Piper Cancer Care-Glendale, Glendale, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Arizona Breast Cancer Specialists-Phoenix, Phoenix, Arizona
  - Arizona Breast Cancer Specialists, Scottsdale, Arizona
  - Arizona Breast Cancer Specialists-Scottsdale, Scottsdale, Arizona
  - Virginia G Piper Cancer Care-Del Camino, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Huntington Memorial Hospital, Pasadena, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Sharp Memorial Hospital, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mills Health Center, San Mateo, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Dominican Santa Cruz Hospital, Santa Cruz, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guiford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - John Fitzgerald Kennedy Medical Center, Atlantis, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Medical Group Urology at Orlando, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Martin Medical Center, Stuart, Florida
  - Robert and Carol Weissman Cancer Center at Martin Health, Stuart, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Elizabeth Health - Lafayette East, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Saint Elizabeth Fort Thomas, Fort Thomas, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Mayo Clinic Radiation Therapy-Northfield, Northfield, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Cancer Partners of Nebraska - Pine Lake, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center - 68th Street Place, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Women's Hospital, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sands Cancer Center, Canandiaqua, New York
  - Putnam Hospital Center, Carmel, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - Vassar Brothers Fishkill Radiation Oncology Center, Fishkill, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Ulster Radiation Oncology Center, Kingston, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Pluta Cancer Center, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Novant Health Breast Surgery - Greensboro, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Novant Health Cancer Institute - Statesville, Stateville, North Carolina
  - NHRMC Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, Wilkesboro, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Wright-Patterson Medical Center, Wpafb, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Evangelical Community Hospital, Lewisburg, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Holy Redeemer Hospital and Medical Center, Meadowbrook, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Radiation Oncology Associates Incorporated, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Lancaster Radiation Therapy Center, Lancaster, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - The West Clinic - Wolf River, Germantown, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Methodist Hospital, Memphis, Tennessee
  - The West Clinic - Mid-Town, Memphis, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Nashville Breast Center, Nashville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology PA Beaumont, Beaumont, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology - Denison Cancer Center, Denison, Texas
  - Texas Oncology-Flower Mound, Flower Mound, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Oncology-Grapevine, Grapevine, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Baylor Medical Center at Irving, Irving, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - MD Anderson League City, League City, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Texas Oncology-McKinney, McKinney, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Scott and White Healthcare Round Rock, Round Rock, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Rutland Regional Medical Center, Rutland, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Sentara Princess Anne Hospital, Virginia Beach, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Tri-Cities Cancer Center, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Seattle Cancer Care Alliance at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Fox Valley Surgical Associates Limited, Appleton, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Regional Medical Center - Appleton, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Surgical Associates of Neenah SC, Neenah, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (14):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-Hopital du Saint-Sacrement (HSS), Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Puerto Rico (4):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Ferrarazzo G, Nieri A, Firpo E, Rattaro A, Mignone A, Guasone F, Manzara A, Perniciaro G, Spinaci S. The Role of Sentinel Lymph Node Biopsy in Breast Cancer Patients Who Become Clinically Node-Negative Following Neo-Adjuvant Chemotherapy: A Literature Review. Curr Oncol. 2023 Sep 25;30(10):8703-8719. doi: 10.3390/curroncol30100630. PMID 37887530
- [Derived] Ditsch N, Rubio IT, Gasparri ML, de Boniface J, Kuehn T. Breast and axillary surgery in malignant breast disease: a review focused on literature of 2018 and 2019. Curr Opin Obstet Gynecol. 2020 Feb;32(1):91-99. doi: 10.1097/GCO.0000000000000593. PMID 31833973
- [Derived] Mamounas ET. Optimal Management of the Axilla: A Look at the Evidence. Adv Surg. 2016 Sep;50(1):29-40. doi: 10.1016/j.yasu.2016.03.003. Epub 2016 Jun 9. No abstract available. PMID 27520860